CLINICAL TRIAL: NCT03748654
Title: Feasibility of Visual Field Testing With a Virtual Reality Headset
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Brennan Eadie (Other)
Responsible Party: Sponsor-Investigator, Brennan Eadie, Assistant Professor, Department of Ophthalmology, Dalhousie University and Nova Scotia Health Authority; MD, PhD, FRCSC, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: E001
Record Dates: First submitted 2018-11-16; First posted 2018-11-21 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Visual Fields

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Patients will perform visual field testing with the Humphrey Field Analyzer and with the Virtual Reality Headset
  Interventions: Diagnostic Test: Visual Field Testing

INTERVENTIONS:
Diagnostic Test: Visual Field Testing — Visual field test using the protocol 24-2 Threshold Test

SUMMARY:
This study aim to determine the feasibility of using a virtual reality (VR) headset (HTC Vive) to test the visual field. The VR headset test will be compared to a conventional visual field test, using the Humphrey Field Analyzer. The investigators will include 10 healthy patients without visual field defect, 10 patients with early glaucomatous visual field defect, and 10 patients with advanced visual field defect. Each patient will perform the conventional test twice and the VR headset test 4 times, divided in 3 visits within a 2 month period. The results of the tests (sensitivity thresholds) will be compared. The investigators hypothesize that the results of the conventional and VR tests will be similar.

ELIGIBILITY:
Inclusion Criteria:

* Previous visual field test with Humphrey Field Analyzer indicating normal field, early glaucomatous field damage, or advanced glaucomatous field damage, according to Canadian Glaucoma Society Guidelines.
* Ability to understand and consent to the study.

Exclusion Criteria:

* Presence of non-glaucomatous pathology that could influence the visual field test, such as media opacities.
* Previous intraocular surgery less than 6 months from inclusion.
* Difficulty to execute a reliable visual field test.
* Potential contra-indications to use of virtual reality headset, including: anxiety disorder, pregnancy, seizure disorder, cardiac pacemaker or other implantable device, severe vertigo or balance disturbance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Visual field differential light sensitivity threshold | Three weeks
  Comparison of differential light sensitivity threshold estimated with the Humphrey Field Analyzer and the Virtual Reality headset

SECONDARY OUTCOMES:
Reproducibility of sensitivity values | Three weeks
  Comparison of the reproducibility of sensitivity values estimated with the Humphrey Field Analyzer and the Virtual Reality headset

CONTACTS AND LOCATIONS:
Overall Officials: Brennan Eadie, MD, PhD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Victoria General Hopsital - Nova Scotia Health Authority, Halifax, Nova Scotia, Canada